CLINICAL TRIAL: NCT03023852
Title: A Phase 1, Open-label, Randomized, Crossover Study in Two Panels of Healthy Adult Subjects to Assess the Relative Oral Bioavailability of a Single Dose of JNJ-63623872/Oseltamivir Fixed-dose Combination Tablet and Single Agent Concept Formulations of JNJ-63623872 Compared to Their Respective Reference Formulation
Brief Title: A Study to Assess the Relative Oral Bioavailability of a Single Dose of JNJ-63623872/Oseltamivir Fixed-dose Combination Tablet and Single Agent Concept Formulations of JNJ-63623872 Compared to Their Respective Reference Formulation in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR108252; 63623872FLZ1011 (Other: Janssen-Cilag International NV); 2016-004504-62 (EudraCT Number)
Record Dates: First submitted 2017-01-16; First posted 2017-01-18 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Healthy
MeSH Terms: interventions — pimodivir; Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Panel 1: Group 1 (Experimental): Participants will receive Treatment A (JNJ-63623872 600 milligram (mg) (2*300 mg) oral tablets [reference]) followed by Treatment B (JNJ- 63623872 600 mg (2*300 mg) concept oral tablet formulation 1 (test 1) and then Treatment C (JNJ-63623872 600 mg (2*300 mg) concept oral tablet formulation 2 (test 2). Each treatment period will be separated 7 days washout period.
  Interventions: Drug: JNJ-63623872
- Panel 1: Group 2 (Experimental): Participants in Group 2 will receive Treatment A followed by Treatment C and then Treatment B with a washout period of minimum 7 days.
  Interventions: Drug: JNJ-63623872
- Panel 1: Group 3 (Experimental): Participants in Group 3 will receive Treatment B followed by Treatment A and then Treatment C with a washout period of minimum 7 days.
  Interventions: Drug: JNJ-63623872
- Panel 1: Group 4 (Experimental): Participants in Group 4 will receive Treatment B followed by Treatment C and then Treatment A with a washout period of minimum 7 days.
  Interventions: Drug: JNJ-63623872
- Panel 1: Group 5 (Experimental): Participants in Group 5 will receive Treatment C followed by Treatment A and then Treatment B with a washout period of minimum 7 days.
  Interventions: Drug: JNJ-63623872
- Panel 1: Group 6 (Experimental): Participants in Group 6 will receive Treatment C followed by Treatment B and then Treatment A with a washout period of minimum 7 days.
  Interventions: Drug: JNJ-63623872
- Panel 2: Group 7 (Experimental): Participants in Group 7 will receive Treatment D [JNJ-63623872/37.5 mg Oseltamivir oral fixed dose combination (FDC) tablet concept formulation (test 3)] followed by Treatment E (JNJ-63623872 600 mg, administered as 2*300 mg and Oseltamivir 75 mg, administered as 1*75 mg). Both treatment periods will be separated with a minimum of 7 days washout period.
  Interventions: Drug: JNJ-63623872; Drug: Oseltamivir
- Panel 2: Group 8 (Experimental): Participants in Group 8 will receive Treatment E followed by Treatment D with a washout period of minimum 7 days.
  Interventions: Drug: JNJ-63623872; Drug: Oseltamivir

INTERVENTIONS:
Drug: JNJ-63623872 — Participants will receive JNJ-63623872 600 mg (2*300 mg) oral tablets in Panel 1 and 2 under Fasted conditions.
Drug: Oseltamivir — Participants will receive Oseltamivir 75 mg (1*75 mg) oral capsule (reference) in Treatment D of Panel 2 and Oseltamivir 75 mg administered as JNJ-63623872/37.5 mg Oseltamivir oral FDC tablet concept formulation (test 3) in Treatment E of Panel 2.
  Arms: Panel 2: Group 7; Panel 2: Group 8

SUMMARY:
The purpose of this study is to assess the rate and extent of absorption of JNJ63623872 following administration of a single oral dose of 2*300 milligram (mg) given as 2 concept single agent tablet formulations compared to the administration of 2*300 mg JNJ63623872 reference tablets, under fasted conditions in healthy adult participants and to assess the rate and extent of absorption of JNJ63623872 and oseltamivir following administration of a single oral dose of 2*300 mg/37.5 mg JNJ63623872/ oseltamivir given as a concept fixed dose combination (FDC) tablet formulation compared to the coadministration of 2*300 mg JNJ63623872 tablets (reference formulation) and 1*75 mg oseltamivir capsule, under fasted conditions in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* A female participant must have a negative serum beta-human chorionic gonadotropin pregnancy test at screening and on Day -1 in each treatment period
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participant participating in clinical studies
* A female participant must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 90 days after receiving the last dose of study drug
* Participant must have a body mass index (BMI), weight kilogram per height square meter square [kg]/height^2 [m]^2) between 18.0 and 30.0 kilogram per meter square (kg/m^2) (extremes included) at screening. The minimum weight will be 50.0 kilogram (kg)
* Participant must have a blood pressure (supine after at least 5 minutes rest) between 90 and 140 millimeters of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic at screening
* Participant must be non-smoker for at least 3 months prior to screening

Exclusion Criteria:

* Participant has history or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders, lipid abnormalities, significant pulmonary disease, diabetes mellitus, hepatic or renal insufficiency, gastrointestinal disease, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participant with a past history of heart arrhythmias (extrasystoli, tachycardia at rest), or history of risk factors for Torsade de Pointes syndrome (eg, hypokalemia, family history of long QT Syndrome)
* Participant with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticaria
* Participant has known allergy to heparin or history of heparin induced thrombocytopenia
* Participant has donated blood or blood products or had substantial loss of blood (more than 500 milliliter (mL) within 3 months before the first administration of study drug or intention to donate blood or blood products during the study
* A woman who is pregnant, or breast-feeding, or planning to become pregnant during this study, or a woman of childbearing potential who is unwilling to use acceptable methods of contraception
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at screening
* Participant has a history of human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection, or tests positive for HIV-1 or -2 at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Predose, 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 48 h, 72 h and 96 hours postdose on Day 5
  The Plasma Concentration (Cmax) is defined as maximum observed plasma concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Predose, 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 48 h, 72 h and 96 hours postdose on Day 5
  The Tmax is defined as actual sampling time to reach maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration Time (AUC [0-Last]) | Predose, 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 48 h, 72 h and 96 hours postdose on Day 5
  AUC last is area under the plasma concentration-time curve from time zero to last quantifiable concentration time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Predose, 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 48 h, 72 h and 96 hours postdose on Day 5
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Apparent Terminal Elimination Rate Constant (Lambda [z]) | Predose, 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 48 h, 72 h and 96 hours postdose on Day 5
  Lambda (z) is defined as apparent terminal elimination rate constant, determined by linear regression using the terminal log-linear phase of the log transformed concentration versus time curve.
Apparent Terminal Elimination Half-life (t1/2) | Predose, 0.5 h, 1 h, 1.5 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 16 h, 24 h, 48 h, 72 h and 96 hours postdose on Day 5
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to follow-up (within 10 to 14 days after last dose)
  Safety and Tolerability
Taste Questionnaire Assessment | Day 1
  A taste questionnaire will be completed by the participants of Panel 2, group 7 within 5 to 15 minutes after intake of the FDC tablet (Treatment E) to evaluate the taste of the oral FDC tablet formulation under fasted conditions. The Taste questionnaire consists of 4 parts (sweetness, bitterness, flavour and overall); each parts is scored on 4 points , i.e. none, weak, moderate and strong.
Swallowability Assessment | Day 1
  Swallowability will be assessed in participants of Panel 2 group 7 on a scale of 1-7; how difficult/easy was it to swallow this tablet. In the scale 0=very difficult and 7=very easy.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- SGS Life Science Services, Antwerp, Belgium